CLINICAL TRIAL: NCT01711424
Title: An Observational Study of OPTIVE PLUS® for the Treatment of Dry Eye Disease
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/DE/012
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-01

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OPTIVE PLUS®: Patients with dry eye prescribed OPTIVE PLUS® in accordance with physician standard practice.
  Interventions: Drug: OPTIVE PLUS®

INTERVENTIONS:
Drug: OPTIVE PLUS® — Patients with dry eye prescribed OPTIVE PLUS® in accordance with physician standard practice.

SUMMARY:
This is an observational study of OPTIVE PLUS® in patients with dry eye disease in a routine clinical setting. Treatment decisions are made by the physician and reflect the physician's current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dry eye
* Physician decision to treat with OPTIVE PLUS® in accordance with the physician's standard practice

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dry eye
Sampling Method: Non-Probability Sample
Enrollment: 1209 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Stuttgart, Baden-Wurttemberg, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients with dry eye prescribed OPTIVE PLUS® in accordance with physician standard practice. There was no investigational drug administered in this study.
Period: Overall Study
Arm/Group | OPTIVE PLUS®
Started | 1209
Completed | 1209
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OPTIVE PLUS®
Number analyzed (Participants) | 1209
Age, Customized [Number; unit: Participants]
  <18 Years | 3 (15.89)
  18 to 30 Years | 51
  31 to 40 Years | 94
  41 to 50 Years | 196
  51 to 60 Years | 230
  61 to 70 Years | 261
  71 to 80 Years | 269
  81 to 90 Years | 84
  >= 91 Years | 5
  Missing data | 16
Sex/Gender, Customized [Number; unit: Participants]
  Male | 398
  Female | 805
  Missing Data | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Very Satisfied or Satisfied With OPTIVE PLUS®
Description: Patients rated their satisfaction with OPTIVE PLUS® as treatment for dry eye signs and symptoms using a 4-point scale (Very satisfied, Satisfied, Dissatisfied or Very dissatisfied).
Time Frame: Week 4
Population: All participants with data available for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | OPTIVE PLUS®
Number analyzed (Participants) | 1191
Participants
  Very satisfied | 356
  Satisfied | 746

2. Secondary Outcome: Number of Participants Where Physician Was Very Satisfied or Satisfied With OPTIVE PLUS®
Description: The physician rated their satisfaction with OPTIVE PLUS® for the treatment of their patient's dry eye signs and symptoms using a 4-point scale (Very satisfied, Satisfied, Dissatisfied or Very dissatisfied).
Time Frame: Week 4
Population: All participants with data available for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | OPTIVE PLUS®
Number analyzed (Participants) | 1176
Participants
  Very satisfied | 367
  Satisfied | 734

3. Secondary Outcome: Tear Break Up Time (TBUT)
Description: TBUT is the time in seconds required for dry spots to appear on the corneal surface after blinking. The longer it takes, the more stable the tear film.
Time Frame: Baseline, Week 4
Population: All participants with complete data available for this outcome measure at Baseline and Week 4.
Measure: Median (Full Range); unit: Seconds
Arm/Group | OPTIVE PLUS®
Number analyzed (Participants) | 475
Seconds
  Baseline | 7.0 [2.0 to 23.0]
  Week 4 | 10.0 [2.0 to 23.0]

4. Secondary Outcome: Schirmer Score
Description: The Schirmer Test measures the rate of the secretion of tears produced by the eye over 5 minutes (min). The results indicate the presence of dry eye (Normal = greater than or equal to 10 millimeters (mm) of tears, Dry Eye = less than 10 mm of tears). The smaller the number, the more severe the dry eye.
Time Frame: Baseline, Week 4
Population: All participants with complete data available for this outcome measure at Baseline and Week 4.
Measure: Median (Full Range); unit: mm/5 min
Arm/Group | OPTIVE PLUS®
Number analyzed (Participants) | 307
mm/5 min
  Baseline | 8.0 [1.0 to 30.0]
  Week 4 | 10.0 [1.0 to 30.0]

ADVERSE EVENTS:
Arm/Group | OPTIVE PLUS®
Serious Adverse Events (participants affected / at risk) | 2/1209
Other Adverse Events (participants affected / at risk) | 0/1209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPTIVE PLUS® (N=1209)
Cataract operation (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.